CLINICAL TRIAL: NCT01175655
Title: A Study to Evaluate the Potential of Mesenchymal Stromal Cells to Treat Obliterative Bronchiolitis After Lung Transplantation
Acronym: MSC in OB
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Prince Charles Hospital (Other Government)
Collaborators: Cell and Tissue Therapies Western Australia (Unknown)
Responsible Party: Principal Investigator, Daniel Chambers, Principal Investigator, The Prince Charles Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC 28105
Record Dates: First submitted 2010-06-25; First posted 2010-08-05 (Estimated); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Bronchiolitis Obliterans; Lung Transplantation
Keywords: Mesenchymal stromal cells; Bronchiolitis obliterans; Lung transplant
MeSH Terms: conditions — Bronchiolitis Obliterans

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MSC (Experimental)
  Interventions: Other: MSC

INTERVENTIONS:
Other: MSC — mesenchymal stromal cells (MSC), aiming for 2 x 106 /kg cells recipient body weight, aiming for a frequency of twice weekly for two weeks

SUMMARY:
The primary aim of this study is to establish the safety of infusions of Mesenchymal Stromal Cells (MSC) from related or unrelated Human Leukocyte Antigen (HLA) identical or HLA mismatched donors in the management of bronchiolitis obliterans syndrome after lung transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with single, bilateral or heart-lung allografts
2. Patients with bronchiolitis obliterans syndrome (BOS) grades 2 & 3 (defined and graded according to international criteria (Appendix 1)), with evidence of deterioration in allograft function (i.e. deteriorating FEV1 or worsening BOS grade) within the last 12 months.
3. Patients with BOS grade 1 and evidence of deterioration in allograft function (i.e. deteriorating FEV1 or worsening BOS grade) within the last 12 months and at least one of the following additional risk factors for subsequent death:

   * Single lung transplant
   * Rapid deterioration (>20% fall in FEV1 in the previous 12 months)
   * A pre-transplant diagnosis of usual interstitial pneumonia (pulmonary fibrosis) or pulmonary hypertension

Exclusion Criteria:

1. Patients with active infection, acute allograft rejection, or airway anastomotic complications
2. Patients with > 3 infective exacerbations of BOS in the last 12 months
3. Patients with a history of cytomegalovirus (CMV) pneumonitis
4. Patients with poor performance status and/or not expected to survive 3 months
5. Patients who are pregnant or breastfeeding
6. Patients with an allergy to beef products.
7. Any condition that in the opinion of the Investigator may interfere with the safety of the patient, his / her completion of required follow-up visits or evaluation of the study objectives.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-02; Primary Completion 2015-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
To establish the safety of infusions of MSC from related or unrelated HLA identical or HLA mismatched donors in the management of bronchiolitis obliterans syndrome after lung transplantation. | 12 months

SECONDARY OUTCOMES:
To document changes in lung function and 6 minute walk distance (6MWD) following infusion of MSC | 12 months
To document survival post MSC infusion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Chambers, A/Prof, Principal Investigator — The Prince Charles Hospital
Locations (2):
- Australia (2):
  - TPCH, Brisbane, Queensland
  - RPH, Perth, Western Australia